CLINICAL TRIAL: NCT01673464
Title: A Prospective Study of Brain Network Activation (BNA) Changes in High School Athletes Following Concussion
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ELM-12
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Mild Traumatic Brain Injury
Keywords: mild Traumatic Brain Injury; mTBI; Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- High School Athletes

SUMMARY:
The main purpose of this study is to prospectively examine changes in Brain Network Activation(BNA)following concussion in high school athletes. In addition, the study will examine the relationship between changes in BNA to symptoms, cognitive performance and vestibular function from baseline to 1-7, 8-14 and 15-21 day post injury intervals in high school athletes with concussion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-18 years
* Able to speak, read and understand English sufficiently to understand the nature of the study, and to allow completion of all study assessments
* Willingness to participate and able to give informed assent (child) and/or consent (parent for minors or adult 18+ years of age for self)

Exclusion Criteria:

* Current or history of TBI (i.e., Glasgow Coma Scale <13) or brain surgery
* Current or history of any psychiatric disorder (except ADD/ADHD), e.g., depression, bipolar disorder, schizophrenic disorder
* Substance abuse within the last year
* Current or history of Special education, e.g., reading disorder (dyslexia), writing disorder (dysgraphia), math disorder (dyscalculia), nonverbal learning disorder
* Current or history of any Neurological disorder, e.g., epilepsy, seizures
* History of any medication affecting CNS within the last year, e.g., antidepressants, anticonvulsants, Ritalin, first generation antihistamines, etc.
* Current or history of Significant sensory deficits such as deafness or blindness
* Current or history of Clinically significant abnormal laboratory values or ECG
* A concussion within the last year
* Current or history of residual symptoms or deficits related to a previous concussion
* Diagnosis of autistic spectrum disorders, e.g., Asperger's syndrome, High functioning Autism, PDD
* Currently with lice or open wounds on scalp
* Long and thick hair that prevents the proper administration of an EEG cap

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: High school (13-18 yrs) athletes from American football, soccer, and lacrosse who meet the inclusion/exclusion criteria will be recruited into the study. We expect that between 10-20 participants will sustain a concussion during the period of the study and complete the post-concussion protocol.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2012-08; Primary Completion 2014-04 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Changes in Brain Network Activation(BNA™)Scores From Baseline Over Post Concussion Recovery Period | baseline, 1-7, 8-14, and 15-21 day post-injury intervals
  To examine prospectively changes in brain network activation (BNA) from baseline to 1-7, 8-14, and 15-21 day post-injury intervals, and/or to recovery (i.e., return to activity) in high school athletes with concussion.

SECONDARY OUTCOMES:
Relationship between changes in BNA to changes in symptoms from baseline over post concussion recovery period | baseline, 1-7, 8-14, and 15-21 day post-injury intervals
  To investigate the relationship between changes in BNA to changes in symptoms from baseline to 1-7, 8-14, and 15-21 day post-injury intervals, and/or to recovery (i.e., return to activity) in high school athletes with concussion.
Relationship between changes in BNA to changes in cognitive performance from baseline over post concussion recovery period | baseline, 1-7, 8-14, and 15-21 day post-injury intervals
  To investigate the relationship between changes in BNA to changes in cognitive performance from baseline to 1-7, 8-14, and 15-21 day post-injury intervals, and/or to recovery (i.e., return to activity) in high school athletes with concussion.
Relationship between changes in BNA to changes in vestibular function from baseline over post concussion recovery period | baseline, 1-7, 8-14, and 15-21 day post-injury intervals
  To investigate the relationship between changes in BNA to changes in vestibular function from baseline to 1-7, 8-14, and 15-21 day post-injury intervals, and/or to recovery (i.e., return to activity) in high school athletes with concussion.

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Sports Medicine Concussion Program, Pittsburgh, Pennsylvania, United States